CLINICAL TRIAL: NCT00852449
Title: Restrictive Versus Liberal Intraoperative Goal-directed Fluid Management During Major Abdominal Surgery:a Prospective Randomized Study
Brief Title: Intraoperative Hypovolemia and Fluid Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple
Other Study IDs: CHU-0045
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Hypovolemia; Organ Dysfunction
Keywords: Intraoperative fluid; Monitoring; Oesophageal Doppler; Abdominal surgery; major abdominal surgery
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- restrictive fluid (Experimental): Restrictive fluid administration: 6 ml kg-1 h-1 of crystalloids (lactated Ringer's solution)
  Interventions: Other: restrictive and liberal fluid therapy
- liberal fluid (Experimental): Liberal fluid administration: 12 ml kg-1 h-1 of crystalloids (lactated Ringer's solution)
  Interventions: Other: restrictive and liberal fluid therapy

INTERVENTIONS:
Other: restrictive and liberal fluid therapy — In both group, when hypovolemia is suspected (peak aortic velocity variation > 13%): fluid bolus (hydroxyethyl starch 130/0.4/6%) according to a predefined algorithm designed to maintain peak aortic velocity < 13% and no further increases in SV

SUMMARY:
Postoperative organ dysfunction severely affects the prognosis of surgical patients. Despite several trials evaluating restrictive or liberal fluid strategies, the ideal fluid replacement strategy remains controversial. Owing to the risk of altered tissue perfusion, a key trigger of organ dysfunction, the purpose of this study was to compare the influence of restrictive and liberal fluid regimens, using a goal-directed approach, on hypovolemia and postoperative organ dysfunction.

DETAILED DESCRIPTION:
Despite several trials evaluating restrictive or liberal fluid strategies, the ideal fluid replacement strategy remains unanswered. Although recent studies suggest that intraoperative fluid restriction may reduce postoperative morbidity and promote faster recovery, extrapolation to individual patients remains difficult. Indeed, whether fluid overload may expose tissue to oedema, impairing oxygenation and wound healing, fluid restriction may, conversely, expose to hypovolemia, which occurs frequently during abdominal surgery, leading to tissue hypoperfusion and organ dysfunction. To date, the restrictive and liberal fluid substitution strategies have not been compared using a goal-directed approach. In addition, recent data suggest that targeting early indicators of hypoperfusion, such as central venous oxygen saturation (ScvO2), which reflects the oxygen delivery/consumption relationship, may be important in the management of patients undergoing major surgery. No data are available on the effects of intraoperative fluid volume replacement strategy on ScvO2 modifications.

The purpose of this study is first to evaluate the influence of restrictive and liberal fluid replacement strategies on both hypovolemia and postoperative organ dysfunction using an oesophageal doppler goal-directed approach (with goal = peak aortic velocity variation and stroke volume optimization) during major abdominal surgery. The second objective is to investigate the effects of fluid loading on ScvO2 modifications.

ELIGIBILITY:
Inclusion Criteria:

* Major intraabdominal surgery

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Body mass index > 35 kg/m2
* Emergency surgery
* Coagulopathy
* Sepsis or Systemic inflammatory response syndrome (SIRS)
* Hepatic failure (prothrombin ratio < 50%, factor V < 50%)
* Contraindication for epidural analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
incidence of intraoperative hypovolemia | intraoperative

SECONDARY OUTCOMES:
postoperative organ failure postoperative complications (included anastomotic leak, perianastomotic abscess) | postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Futier, Principal Investigator — University Hospital, Clermont-Ferrand

REFERENCES:
- [Derived] Futier E, Constantin JM, Petit A, Chanques G, Kwiatkowski F, Flamein R, Slim K, Sapin V, Jaber S, Bazin JE. Conservative vs restrictive individualized goal-directed fluid replacement strategy in major abdominal surgery: A prospective randomized trial. Arch Surg. 2010 Dec;145(12):1193-200. doi: 10.1001/archsurg.2010.275. PMID 21173294
- [Derived] Futier E, Robin E, Jabaudon M, Guerin R, Petit A, Bazin JE, Constantin JM, Vallet B. Central venous O(2) saturation and venous-to-arterial CO(2) difference as complementary tools for goal-directed therapy during high-risk surgery. Crit Care. 2010;14(5):R193. doi: 10.1186/cc9310. Epub 2010 Oct 29. PMID 21034476